CLINICAL TRIAL: NCT07400952
Title: Multicenter, Randomized, Double-Masked, Placebo-Controlled Study to Evaluate the Safety and Efficacy of GLK-221 Ophthalmic Solution in Subjects With Keratoconus
Brief Title: Placebo-controlled Study to Evaluate the Safety and Efficacy of GLK-221 Ophthalmic Solution in Subjects With Keratoconus
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Glaukos Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GLK-221-01
Record Dates: First submitted 2026-02-03; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Keratoconus
Keywords: Keratoconus
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- GLK-221 Ophthalmic Solution (Experimental): GLK-221 Ophthalmic Solution administered topically twice daily to both eyes
  Interventions: Drug: GLK-221 Ophthalmic Solution
- Placebo (Placebo Comparator): Placebo Ophthalmic Solution administered topically twice daily to both eyes
  Interventions: Drug: Placebo Ophthalmic Solution

INTERVENTIONS:
Drug: GLK-221 Ophthalmic Solution — GLK-221 Ophthalmic Solution administered twice daily to both eyes
  Arms: GLK-221 Ophthalmic Solution
Drug: Placebo Ophthalmic Solution — Placebo Ophthalmic Solution administered twice daily to both eyes
  Arms: Placebo

SUMMARY:
Multi-center, parallel-group, placebo-controlled trial designed to assess the safety and efficacy of twice-daily topically administered GLK-221 Ophthalmic Solution in subjects with keratoconus.

ELIGIBILITY:
Inclusion Criteria:

* Be ≥ 18 and ≤ 55 years of age
* Diagnosis of keratoconus in the study eye

Exclusion Criteria:

* Pregnant, lactating or planning a pregnancy
* Currently enrolled, or within 30 days prior to Screening were enrolled, in another investigational drug or device trial

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-12-23 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Mean change from baseline in maximum corneal curvature | 16 weeks
  Mean change from baseline in maximum corneal curvature

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, MD, Study Director — Glaukos Corporation
Locations (1):
- Glaukos Clinical Study Site, Westerville, Ohio, United States

IPD SHARING:
Plan to Share IPD: No